CLINICAL TRIAL: NCT04937946
Title: Efficacy and Safety of Fentanyl for Pain Control in Newborns on Mechanical Ventilation
Brief Title: Efficacy and Safety of Fentanyl for Pain Control in Newborn on Mechanical Ventilation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Kundan Kumar Yadav, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3491
Record Dates: First submitted 2021-06-19; First posted 2021-06-24 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Mechanical Ventilation Complication
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fentanyl (Experimental): Fentanyl will be given within 24 hours from the initiation of mechanical ventilation at an intravenous loading dose of 1 microgram/kg in 30 minutes, followed by a continuous intravenous infusion of 1μg/kg/hour up to 5 days or until the end of mechanical ventilation (if interrupted before 5 days ).
  Interventions: Drug: Fentanyl
- Placebo (No Intervention): Will receive continuous infusion of IV fluid up to 5 days or until the end of mechanical ventilation (if interrupted before 5 days ).

INTERVENTIONS:
Drug: Fentanyl — Fentanyl will be administered as an intravenous loading dose of 1 microgram/kg in 30 minutes, followed by a continuous intravenous infusion of 1μg/kg/hour. The infusion will be administered through a peripheral line. Fentanyl infusion will be initiated within 24 hours after the start of mechanical ventilation and will be continued until the end of mechanical ventilation, and not longer than 5 days .
  Arms: Fentanyl

SUMMARY:
The purpose of the study is to assess the efficacy and safety of Fentanyl for pain control in Newborns on mechanical ventilator.

DETAILED DESCRIPTION:
This Randomized Controlled Trial will be conducted in the Department of Neonatology, BSMMU, Dhaka after approval by Institutional Review Board (IRB). A Written informed consent will be obtained before enrollment in the study from the parents or guardians. . The study cohort will comprise all inborn and outborn newborns admitted to the neonatal intensive care unit (NICU) who receive mechanical ventilation administered through an endotracheal tube . The enrolled neonates will be randomly assigned with computer-generated random number tables via software named 'Random Allocation Software', to receive either of the intervention.

Once the parents will agree to the study and provide signed informed consent, all eligible neonates will be randomized to start treatment within 24 hours from the initiation of mechanical ventilation. Randomized infants will be allocated to the fentanyl group to receive a continuous infusion of fentanyl or to the placebo group to receive a continuous infusion of iv fluid.

Fentanyl will be administered as an intravenous loading dose of 1 microgram/kg in 30 minutes, followed by a continuous intravenous infusion of 1μg/kg/hour. The infusion will be administered through a peripheral line. Fentanyl infusion will be initiated within 24 hours after the start of mechanical ventilation and will be continued until the end of mechanical ventilation, and not longer than 5 days .

ELIGIBILITY:
Inclusion Criteria:

1. All inborn and outborn newborns admitted to the neonatal intensive care unit (NICU) who received mechanical ventilation administered through an endotracheal tube.
2. Newborn on mechanical ventilator for at least 72 hours.

Exclusion Criteria:

1. Known genetic or chromosomal disorders,
2. The need for postoperative analgesic therapy during the study period,
3. Major congenital anomaly,
4. Those who received drugs like midazolam, paracetamol, morphine, muscle relaxants, phenobarbital, phenytoin, and chloral hydrate during the study period.
5. Probable rapid extubation.

Ages: 1 Hour to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Decrease in Neonatal Pain Agitation and Sedation Scale (NPASS) score. | 5 days
  If fentanyl is able to decrease NPASS pain score. Total score is 13. A mean difference of 3 points will be considered clinically relevant.

SECONDARY OUTCOMES:
Adverse effects of fentanyl | 5 days
  Duration of mechanical ventilation (hours); chest wall rigidity (evaluated by clinical observation), diuresis, hypotension

CONTACTS AND LOCATIONS:
Overall Officials: BSMMU, Study Chair — Bngabandhu Sheikh Mujib Medical University

IPD SHARING:
Plan to Share IPD: Yes
After the approval of Institutional Review Board
Time Frame: August 2021 to July 2022
Access Criteria: After the approval of Institutional Review Board